CLINICAL TRIAL: NCT02836795
Title: A Phase I, Open Label, Single Center and Dose Escalation Study Investigating Tolerance and Pharmacokinetics of Single and Multiple Doses of Recombinant Humanized Anti-PD-1 Monoclonal Antibody for Injection in Patients With Advanced Solid Tumors
Brief Title: Safety and Tolerability of Recombinant Humanized Anti-PD-1 Monoclonal Antibody Toripalimab for Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Junshi-JS001-BJZL-I
Record Dates: First submitted 2016-07-11; First posted 2016-07-19 (Estimated); Last update posted 2025-06-08 (Actual); Status verified 2019-10

CONDITIONS: Melanoma; Urological Cancer
Keywords: anti-PD-1 monoclonal antibody; advanced solid tumors; safety
MeSH Terms: conditions — Melanoma; Urologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- humanized anti-PD-1 monoclonal antibody Toripalimab (Experimental): humanized anti-PD-1 monoclonal antibody is to be injected intravenously 1mg/kg or 3mg/kg or 10mg/kg until disease progresses or unacceptable tolerability occurs.
  Interventions: Biological: humanized anti-PD-1 monoclonal antibody Toripalimab (JS001)

INTERVENTIONS:
Biological: humanized anti-PD-1 monoclonal antibody Toripalimab (JS001) — humanized anti-PD-1 monoclonal antibody (JS001) is a programmed death-1 (PD-1) immune checkpoint inhibitor antibody, which selectively interferes with the combination of PD-1 with its ligands, PD-L1 and PD-L2, resulting in the activation of lymphocytes and elimination of malignancy theoretically.
  Other Names: JS001, TAB001

SUMMARY:
This is a mono-center, open-label, phase 1 study evaluating the humanized anti-PD-1 antibody JS001, as a monotherapy in patients with advanced melanoma or urological cancers who have failed in routine systemic treatment. The study will be conducted in 2 parts: dose escalation and cohort expansion to investigate tolerability and efficacy.

DETAILED DESCRIPTION:
This is a mono-center, open-label, phase 1 study evaluating the humanized anti-PD-1 antibody JS001, as a monotherapy in patients with advanced solid tumor (melanoma or urological cancers) who have failed in previous routine systemic treatment. The study will be conducted in 2 parts: dose escalation and cohort expansion. In the first part, nine patients are injected with different dosage of the humanized anti-PD-1 antibody (1mg/kg or 3mg/kg or 10mg/mg, three patients in one group ) once and observed carefully in the following 4 weeks. If no dose-limiting toxicity (DLT) occurs, then they are injected every 2 weeks until disease progresses or unacceptable toxicity occurs. This part is to confirm DLT, maximum tolerated dose (MTD) and recommended dose (RD). In the second part, 6-12 patients are enrolled in each dosage group and injected with the humanized anti-PD-1 antibody every 2 weeks until disease progresses or unacceptable toxicity occurs. This part is to further analyze safety and efficacy of the humanized anti-PD-1 antibody.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female aged 18 to 70 years are eligible;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Histologic diagnosis of unresectable melanoma or urological cancer. Have failed at least 1 prior routine regimen for metastatic disease, or failed to tolerate the toxicity, or lack of any routine regimens.
* Providing with tumor specimen (for testing the expression of PD -L1 and the infiltrating lymphocytes);
* At least 1 measurable lesion (only 1 measurable lymph node lesion is excluded) (routine CT scan >=20mm, spiral CT scan >=10mm, no prior radiation to measurable lesions) Predicted survival >=6 months;
* Brain or meningeal metastases must be disposed with surgery or radiation, and be stable clinically for at least 8 weeks (prior systemic steroids was allowed, but concurrent administration of systemic steroids with the study drug is excluded).
* Screening laboratory values must meet the following criteria（within past 14 days）:

hemoglobin ≥ 9.0 g/dL neutrophils ≥ 1500 cells/ µL platelets ≥ 100 x 10^3/ µL total bilirubin ≤ 1.5 x upper limit of normal (ULN) aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis serum creatinine ≤1╳ULN，creatinine clearance >50ml/min (Cockcroft-Gault equation)

* Without systemic steroids within past 4 weeks
* Males or female of childbearing potential must: agree to use using a reliable form of contraception (eg, oral contraceptives, intrauterine device, control sex desire, double barrier method of condom and spermicidal) during the treatment period and for at least 12 months after the last dose of study drug.
* Must have read, understood, and provided written informed consent voluntarily. Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Hypersensitivity to recombinant humanized anti-PD-1 monoclonal Ab or its components.
* Prior treatment with mAb within past 3 months (locally administration excluded)
* Prior antitumor therapy (including corticosteroids and immunotherapy) or participation in other clinical trials within past 4 weeks, or have not recovered from toxicities since the last treatment;
* Pregnant or nursing
* Abnormal Blood coagulation
* Positive tests for HIV, HCV, HBsAg or HBcAb with positive test for HBV DNA (>500IU/ml)
* History with pulmonary tuberculosis;
* Patients with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism or hypothyroidism.
* Severe, uncontrolled medical condition that would affect patients' compliance or obscure the interpretation of toxicity determination or adverse events, including active severe infection, uncontrolled diabetes, angiocardiopathy (heart failure > class II NYHA, heart block >II grade, myocardial infarction, unstable arrhythmia or unstable angina within past 6 months, cerebral infarction within past 3 months) or pulmonary disease ( interstitial pneumonia, obstructive pulmonary disease or symptomatic bronchospasm).
* Evidence with CNS disease.
* Prior treatment with bone marrow stimulating factors，such as CSF (colony stimulating factor), EPO (erythropoietin), within past 1 weeks
* Prior live vaccine therapy within past 4 weeks.
* Prior major surgery within past 4 weeks (diagnostic surgery excluded).
* Psychiatric medicines abuse without withdrawal, or history of psychiatric illness.
* Prior malignancy active within the previous 5 years except for locally curable cancers that have been apparently cured, such as basal cell skin cancer or carcinoma in situ of the cervix.
* Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1.5 years

SECONDARY OUTCOMES:
PD-1 receptor occupancy of blood | 1.5 years
Objective Response Rate (ORR) by irRC and RECIST 1.1 | 3 years
Duration of Response (DOR) by irRC and RECIST 1.1 | 3 years
Disease Control Rate (DCR) by irRC and RECIST 1.1 | 3 year
Time to response (TTR) by irRC and RECIST 1.1 | 3 years
Progression-free survival(PFS) by irRC and RECIST 1.1 | 3 years
Overall survival (OS) by irRC and RECIST 1.1 | 3 years
Maximum Plasma Concentration (Cmax) after single dose injection of Anti-PD-1 Monoclonal Antibody (mAb) | 1.5 years
Peak Time (Tmax) after single dose injection of Anti-PD-1 mAb | 1.5 years
Area Under the Curve (AUC) after single dose injection of Anti-PD-1 mAb | 1.5 years
t1/2 after single dose injection of Recombinant Humanized Anti-PD-1 mAb | 1.5 years
Plasma clearance (CL) after single dose injection of Anti-PD-1 mAb | 1.5 years
Apparent volume of distribution (V) after single dose injection of Anti-PD-1 mAb | 1.5 years
Minimum Plasma Concentration (Cmin) of steady state after multiple dose injection of Anti-PD-1 mAb | 1.5 years
Average Plasma Concentration (Cav) of steady state after multiple dose injection of Anti-PD-1 mAb | 1.5 years
degree of fluctuation (DF) of steady state after multiple dose injection of Anti-PD-1 mAb | 1.5 years
Apparent volume of distribution of steady state (Vss) after multiple dose injection of Anti-PD-1 mAb | 1.5 years

OTHER OUTCOMES:
correlation analysis of PD-L1 expression of tumor and ORR | 3 years
correlation analysis of PD-L1 expression of tumor and DOR | 3 years
correlation analysis of PD-L1 expression of tumor and DCR | 3 years
correlation analysis of PD-L1 expression of tumor and TTR | 3 years
correlation analysis of PD-L1 expression of tumor and PFS | 3 years
correlation analysis of PD-L1 expression of tumor and OS | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Phd MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chen R, Peng PC, Wen B, Li FY, Xie S, Chen G, Lu J, Peng Z, Tang SB, Liang YM, Deng X. Anti-Programmed Cell Death (PD)-1 Immunotherapy for Malignant Tumor: A Systematic Review and Meta-Analysis. Transl Oncol. 2016 Feb;9(1):32-40. doi: 10.1016/j.tranon.2015.11.010. PMID 26947879
- [Background] Ribas A, Puzanov I, Dummer R, Schadendorf D, Hamid O, Robert C, Hodi FS, Schachter J, Pavlick AC, Lewis KD, Cranmer LD, Blank CU, O'Day SJ, Ascierto PA, Salama AK, Margolin KA, Loquai C, Eigentler TK, Gangadhar TC, Carlino MS, Agarwala SS, Moschos SJ, Sosman JA, Goldinger SM, Shapira-Frommer R, Gonzalez R, Kirkwood JM, Wolchok JD, Eggermont A, Li XN, Zhou W, Zernhelt AM, Lis J, Ebbinghaus S, Kang SP, Daud A. Pembrolizumab versus investigator-choice chemotherapy for ipilimumab-refractory melanoma (KEYNOTE-002): a randomised, controlled, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):908-18. doi: 10.1016/S1470-2045(15)00083-2. Epub 2015 Jun 23. PMID 26115796
- [Derived] Tang B, Yan X, Sheng X, Si L, Cui C, Kong Y, Mao L, Lian B, Bai X, Wang X, Li S, Zhou L, Yu J, Dai J, Wang K, Hu J, Dong L, Song H, Wu H, Feng H, Yao S, Chi Z, Guo J. Safety and clinical activity with an anti-PD-1 antibody JS001 in advanced melanoma or urologic cancer patients. J Hematol Oncol. 2019 Jan 14;12(1):7. doi: 10.1186/s13045-018-0693-2. PMID 30642373